CLINICAL TRIAL: NCT07153627
Title: Rectal Ozone as Neuroprotector Post CNS Insult in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abd ELgawad Mohamed Asfour, Assistant Lecturer of Pediatrics, Faculty of Medicine, Al-Azhar University, Egypt., Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-623
Record Dates: First submitted 2025-08-19; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Rectal Ozone; Neuroprotector; CNS; Insult; Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients will receive 40 Rectal ozone sessions or until improvement (maximum 80 sessions), in addition to their conventional rehabilitation program.
  Interventions: Other: Rectal ozone sessions
- Group 2 (Active Comparator): Patients will receive their conventional rehabilitation program only (physiotherapy sessions three times per week for the treatment period (six months).
  Interventions: Other: Conventional rehabilitation program

INTERVENTIONS:
Other: Rectal ozone sessions — Patients will receive 40 Rectal ozone sessions or until improvement (maximum 80 sessions), in addition to their conventional rehabilitation program.
  Arms: Group I
Other: Conventional rehabilitation program — Patients will receive their conventional rehabilitation program only (physiotherapy sessions three times per week for the treatment period (six months).
  Arms: Group 2

SUMMARY:
This study aims to evaluate the efficacy of rectal ozone therapy as a neuroprotective modality in Pediatric acquired brain injury.

DETAILED DESCRIPTION:
Acquired brain injury (ABI) from primary neurologic diagnoses accounts for 20% of all pediatric critical care admissions and more than 60,000 hospital admissions annually.

Ozone (O3) gas was discovered in the 1840s, and soon after that, the scientific community began to expand past the notion that it was just another gas of the Earth's atmosphere.

ELIGIBILITY:
Inclusion Criteria:

* Age from 1 month to 18 years.
* Both sexes.
* Children admitted to the pediatric intensive care unit (PICU) with acquired neurological insult.
* Children with neurological sequelae
* Children who are exposed to acquired brain injury, e.g., traumatic brain injury, cardiac arrest, intracranial hemorrhage, central nervous system infections, stroke, tumor, or hypoxia, with neurological sequelae diagnosed by neurological examination and magnetic resonance imaging (MRI), to detect that disorder early.

Exclusion Criteria:

* Patients with no degree of disability or sequelae.
* Patients not fit for Rectal ozone therapy.
* Patients with active epilepsy and recurrent seizures.
* Children with a positive family history of degenerative brain insults.
* Children with behavioral problems.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of muscle Tone | 6 months post-sessions
  Assessment of muscle tone (degree of spasticity) of affected child according to Modified Ashworth's Scale. Ashworth's scale is a 6-point scale, from 0 to 4, with higher scores indicating greater spasticity.

SECONDARY OUTCOMES:
Incidence of reduction in neuroinflammation | 6 months post-sessions
  Incidence of reduction in neuroinflammation will be recorded.
Assessment of quality of life | 6 months post-sessions
  Assessment of quality of life including emotional well-being or social interaction will be recorded.
Incidence of adverse effects | 6 months post-sessions
  Incidence of adverse effects will be recorded.
Measurement of age-related response variability | 6 months post-sessions
  Age-related response variability by evaluating how different age groups respond to treatment will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.